CLINICAL TRIAL: NCT06116305
Title: Lactate Kinetics as a Predictor of Survival in ACLF With Septic Shock: A Prospective Observational Study
Brief Title: Lactate Kinetics as a Predictor of Survival in ACLF With Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-ACLF-13
Record Dates: First submitted 2023-09-29; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-09

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Shock is a clinical state of tissue hypoxia. This hypoxia may be brought about by either decreased perfusion or the inability of the cell to extract oxygen in the presence of adequate perfusion. This causes cellular dysfunction. The most encountered form of shock seen in cirrhotics is septic shock. Septic shock has underlying cellular and metabolic abnormalities in addition to circulatory dysfunction. The circulatory dysfunction in sepsis is in the form of severe vasodilatation with high cardiac index. Cirrhosis is a state of hyperdynamic circulation. The mortality of septic shock in these group of patients is still higher. Sepsis-3 definition of septic shock describes it as a dysregulated immune response to an infection, leading to systemic inflammation, vasodilation, and organ impairment (3). Practically, to define septic shock it requires the lactate to be more than 2 mmol/L and there should be requirement of vasopressors after adequate fluid resuscitation.

Increased lactate levels can indicate tissue hypoxia, excessively rapid aerobic glycolysis, or reduced clearance. As lactate is a normal product of glucose and pyruvate metabolism, any increase in glucose metabolism and / or decrease in pyruvate metabolism will increase lactate generation. This was observed even in the presence of adequate tissue oxygenation. In sepsis, the inflammatory response appears to be associated with an increase in glycolysis and impaired pyruvate dehydrogenase activity. Thus, cytoplasmic pyruvate increases with greater lactate formation. The glycolytic enzyme complex lactate dehydrogenase (LDH) regenerates nicotinamide adenine dinucleotide (NAD) when pyruvate is reduced to lactate via a redox-coupled process in anaerobic glycolysis (Embden-Meyerhof pathway). Since lactate is overproduced and underutilised in tissue hypoxia due to poor mitochondrial oxidation, lactate has traditionally been used as a diagnostic marker for tissue hypoxia. However, up to 70% of the body's lactate elimination occurs in the liver

DETAILED DESCRIPTION:
• We hypothesise that delta lactate at 6 hours would be a better predictor of survival in patients of ACLF with septic shock when compared to admission lactate

Aim and Objective -

* Aim: To study the impact of measurement of dynamic change of lactate on outcomes in ACLF patients with septic shock
* Primary objective: Delta arterial lactate at 6 hours (delta lactate) as a predictor of survival at 7 days in patients of ACLF with septic shock

Secondary objectives:

* To study the lactate kinetics and lactate clearance at different time points (0, 6, 12,24,48 and 72 hours)
* Impact of delta arterial lactate and lactate clearance at 6h on the length of hospital stay, days of ventilation, time taken for reversal of shock and 28-day mortality
* Impact of oxygenation, respiratory acidosis, metabolic acidosis, anion gap
* Effect of etiology of ACLF on lactate kinetics
* Study the impact of type of infection (MDRO) on lactate kinetics
* Study the impact of therapeutic interventions ( CRRT - impact of CRRT in a subgroup / Fluids/ Vasopressors) on lactate kinetics in ACLF patients with septic shock at day 7
* To develop a dynamic predictive model incorporating lactate kinetics to improve risk stratification and prediction of 28-day mortality.

Methodology:

Study population: Patients of ACLF with septic shock who get admitted to our ICU with a diagnosis of septic shock in the age group 18 - 70 years.

Study design: Prospective observational study Study period: 3 months

Study Location: Department of Hepatology, ILBS, New Delhi

Definitions Sepsis will be defined as a SOFA score more than 2 (or increase in SOFA score >2) in a patient with a suspected infection

Septic shock will be defined as Subset of patients with sepsis with hypotension (MAP <65) unresponsive to fluid boluses AND with lactate >2mmol/L despite adequate fluid resuscitation

Reversal of Shock will be defined as maintenance of MAP > 65mmHg after discontinuation of all vasopressors for 6 hours.

Lactic Acidosis

Hyperlactatemia

* Sample size with justification: No study has been done on lactate clearance in ACLF (APASL) with septic shock
* We have taken a sample size of 100 arbitrarily

  * Intervention: Not applicable (Observational study)
  * Monitoring and assessment:
  * Statistical Analysis: Continuous data- Student's t test
  * Nonparametric analysis- Mann Whitney test
  * Survival outcome By Kaplan-Meier method curve.
  * For all tests, p≤ 0.05 will be considered statistically significant.
  * Analysis will be performed using SPSS .
  * The analysis will be done with intention to treat and per protocol analysis if
  * Adverse effects: N/A
  * Stopping rule of study: N/A

ELIGIBILITY:
Inclusion Criteria:

1. Patients of Acute on chronic liver failure with septic shock (APASL, Sepsis -3 definitions)
2. Age 18-70yrs
3. Informed Consent

Exclusion Criteria:

1. Acute coronary syndrome, hemodynamically unstable arrhythmias
2. CKD stage 5
3. COPD with acute exacerbation
4. Acute CVA or Seizures
5. Extremely moribund patients
6. Hepato-cellular carcinoma (HCC), intrahepatic or extrahepatic malignancy
7. Pregnancy
8. Diabetic ketoacidosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of ACLF with septic shock who get admitted to our ICU with a diagnosis of septic shock in the age group 18 - 70 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-05 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants survived at day 7 | 7 days

SECONDARY OUTCOMES:
lactate clearance and delta lactate will be measured --> lactate clearance = (Initial lactate - current lactate) Initial lactate * 100, Delta lactate = Initial lactate - current lactate | 0 hours
lactate clearance and delta lactate will be measured --> lactate clearance = (Initial lactate - current lactate) Initial lactate * 100, Delta lactate = Initial lactate - current lactate | 6 hours
lactate clearance and delta lactate will be measured --> lactate clearance = (Initial lactate - current lactate) Initial lactate * 100, Delta lactate = Initial lactate - current lactate | 12 hours
lactate clearance and delta lactate will be measured --> lactate clearance = (Initial lactate - current lactate) Initial lactate * 100, Delta lactate = Initial lactate - current lactate | 24 hours
lactate clearance and delta lactate will be measured --> lactate clearance = (Initial lactate - current lactate) Initial lactate * 100, Delta lactate = Initial lactate - current lactate | 48 hours
lactate clearance and delta lactate will be measured --> lactate clearance = (Initial lactate - current lactate) Initial lactate * 100, Delta lactate = Initial lactate - current lactate | 72 hours
Impact of delta arterial lactate at 6 hours on length of hospital stay (measured in days). | 28 days
Impact of delta arterial lactate at 6 hours on need of invasive ventillation (Yes/no) | 7 days
Impact of delta arterial lactate at 6 hours on number of days of invasive ventillation (Measured in days) | 7 days
Impact of lactate clearance at 6 hours on length of hospital stay (measured in days). | 28 days
impact of lactate clearance at 6 hrs on need of invasive ventillation (Yes/no), | 7 days
impact of lactate clearance at 6 hrs on number of days of invasive ventillation (Measured in days) | 7 days
Length of hospital stay (measured in days). | 28 days
Need of ventilation | 28 days
Days of ventilation | 28 days
impact of oxygenation measured by PF ratio at 0H on delta lactate at 6 hours | 6 hours
Correlation between presence or absence of metabolic acidosis with delta lactate at 6 hours | 6 hours
Number of patients with effect of anion gap at 0H if metabolic acidosis is present on the delta lactate at 6 hours | 6 hours
Number of patients with effect of ejection fraction / cardiac outout on delta arterial lactate at 6 hours | 6 hours
To study the impact of presence or absence of multi drug resistant organism (in culture or PCR anallysis) on delta lactate at 6 hours | 7 days
The effect of need of renal replacement therapy (till day 7) on delta lactate at 6 hours | 7 days
The effect of number of days of continuous renal replacement therapy (till day7) on delta lactate at 6 hours | 7 days
The amount of fluid resuscitated and its effect on delta lactate at 6 hours | 7 days
Number of patients with number of patients with Noradrenaline requirement and effect on delta lactate at 6 hours | 7 days
To study the effect of lactate kinetics on 28 day mortality and to study the other factors affecting 28 day mortality | 28 days
Coerrelation between presence or absence of respiratory acidosis on the delta lactate at 6 hours | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided